CLINICAL TRIAL: NCT00554983
Title: A Multicentre Randomised Placebo-controlled Double-blind Pivotal Clinical Trial for the Evaluation of Safety and Efficacy of Specific Immunotherapy With an Aluminium Hydroxide-adsorbed Recombinant Hypoallergenic Derivative of the Major Birch Pollen Allergen, rBet v 1-FV
Brief Title: Efficacy and Safety From a Recombinant Folding Variant of Bet v 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AL0702rB; 2007-001029-84 (EudraCT Number)
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Allergy
Keywords: Recombinant birch pollen allergy; IgE-mediated allergic disease attributed to birch pollen
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator)
  Interventions: Biological: placebo
- 1 (Experimental)
  Interventions: Biological: recombinant birch pollen allergen

INTERVENTIONS:
Biological: recombinant birch pollen allergen — subcutaneous injections (s.c.). Dosage escalation phase from 0.75 to 80 microgram maintenance dose s.c. injections of 80 microgram
  Arms: 1
Biological: placebo — subcutaneous injections (s.c.). Dosage escalation phase from 0.75 to 80 microgram maintenance dose s.c. injections of 80 microgram
  Arms: 2

SUMMARY:
Efficacy and Safety from a recombinant folding variant of Bet v 1

ELIGIBILITY:
Inclusion Criteria:

* Allergic rhinoconjunctivitis attributable to birch pollen
* Positive SPT
* Positive EAST
* Positive specific provocation test

Exclusion Criteria:

* Serious chronic diseases
* Other perennial allergies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 255 (Actual)
Dates: Start 2007-09; Primary Completion 2010-06 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Symptom-Medication-Score | during pollen season

CONTACTS AND LOCATIONS:
Overall Officials: Ludger Klimek, Professor, Principal Investigator
Locations (1):
- Allergopharma GmbH & Co. KG, Reinbek, Germany

REFERENCES:
- See also: Leader in specific allergy research and therapy — http://www.allergopharma.de
- See also: Click here for information about this trial in the European Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/trial/2007-001029-84/DE